CLINICAL TRIAL: NCT02295215
Title: Effects of Physical Training on Sensitivity Baroreflex Patients Without Chagas' Heart Ventricular Systolic Dysfunction
Brief Title: Exercise Training in Patients With Chagasic Heart Disease Without Ventricular Dysfunction
Acronym: CH0660/10
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT01900000
Record Dates: First submitted 2014-08-25; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2013-06

CONDITIONS: Chagas Disease
Keywords: chagas disease; exercise; baroreflex sensitivity
MeSH Terms: conditions — Chagas Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedentary Group (No Intervention): The patients will not do exercise training
- Trained Group (Experimental): The patients will do exercise training for sixteen weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise Training for 4 months
  Arms: Trained Group

SUMMARY:
The prevalence of Chagas' disease continues high even in the developed countries. Chagasic Cardiomyopathy with preserved ventricular function is an understudied form of Chagas disease. Since a majority of patients with these changes progress to dilated form with ventricular dysfunction with all its serious consequences, it is interesting to better understand the pathophysiology of the disease at the stage where there electrocardiographic changes and preserved ventricular function. And besides, search strategies to slow the progress, or even prevent the chronic phase of the disease. For this reason the investigators will evaluate the effects of exercise training in patients with Chagas cardiomyopathy without ventricular dysfunction.

DETAILED DESCRIPTION:
Chagasic Cardiomyopathy with preserved ventricular function is an understudied form of Chagas disease. Since a majority of patients with these changes progress to dilated form with ventricular dysfunction with all its serious consequences, it is interesting to better understand the pathophysiology of the disease at the stage where there electrocardiographic changes and preserved ventricular function. And besides, search strategies to slow the progress, or even prevent the chronic phase of the disease. For this reason the investigators will evaluate the effects of exercise training in patients with Chagas cardiomyopathy without ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Chagas' disease patients, diagnosed with at least two positive serological reactions to Chagas' disease,
* Ejection fraction ≥55%

Exclusion Criteria:

* Participation in a regular exercise program in the last 3 months preceding the survey
* Use of oral anticoagulant
* Use of a pacemaker or implantable cardioverter
* Hemodynamic instability
* Myocardial revascularization infarction or unstable angina in the last 3 months of the start of the protocol
* Diabetes mellitus
* Hypertension
* Pulmonary Disease
* Valvular lesions
* Atrial Fibrillation
* Angina of effort

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Sympathetic nerve activityAutonomic control | 4 months
  Exercise training will improve baroreflex sensitivity and reduce sympathetic nerve activity.

SECONDARY OUTCOMES:
Peak oxygen consumption | 4 months
  Exercise training will improve peak oxygen consumption
Skeletal muscle strength | 4 months
  Exercise training will increase skeletal muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Adriana O Sarmento, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Heart Institute - HC-FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Sarmento AO, Antunes-Correa LM, Alves MJNN, Bacurau AVN, Fonseca KCB, Pessoa FG, Lobo DML, Moreira LDP, Trombetta IC, Rondon MUPB, Rondon E, Vieira MLC, Ramires FJA, do Brasileiro-Santos MS, Brum PC, Mady C, Negrao CE, Thomas S, Ianni BM. Effect of exercise training on cardiovascular autonomic and muscular function in subclinical Chagas cardiomyopathy: a randomized controlled trial. Clin Auton Res. 2021 Apr;31(2):239-251. doi: 10.1007/s10286-020-00721-1. Epub 2020 Sep 1. PMID 32875456